CLINICAL TRIAL: NCT03697044
Title: Irinotecan Loaded Drug-eluting Beads (DEBIRI) for the Treatment of Liver Metastases From Colorectal Cancer - An Observational Study and Patient Registry
Brief Title: Irinotecan Drug-eluting Bead Liver Embolisation Registry
Acronym: DLivERDEBIRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Damian Mullan, Consultant Radiologist, The Christie NHS Foundation Trust
Other Study IDs: Christie NHS
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Irinotecan Drug-Eluting-Bead Trans Arterial ChemoEmbolisation — Patient Registry to assess the delivery of Irinotecan loaded drug eluting beads for the treatment of colorectal liver cancer metastases.
  Other Names: DEBIRI; DEB TACE

SUMMARY:
Purpose:

The purpose of this study is: to assess and define the current practice of the delivery of irinotecan loaded drug eluting beads in the treatment of liver metastases from colorectal cancer; to correlate how the delivery of this drug compares to worldwide/European guidelines, and to determine which individual variations in delivery may be associated with an increased complication profile or better outcome.

The aim of the study is to:

1. Prospectively evaluate the number of centres providing DEBIRI
2. To determine the number of patients being treated nationally per year
3. To evaluate individual variations in practice with respect to number of treatments, method of pain control, side effect profile, and complication profile.
4. To collect patient specific data subsets to allow correlation and causal associations between these individual variations, and relate these to efficacy and survival during the study period.

DETAILED DESCRIPTION:
The study is to evaluate and audit the use of drug eluting beads loaded with irinotecan chemotherapy for the treatment of colorectal liver metastases. Colorectal cancer (CRC) is the third most common malignancy in men and the second in women, affecting more than 1.2 million people per year worldwide.

The development of metastases is the main cause of death in patients with CRC. Surgical resection is the first-line treatment for hepatic CRC metastases.

Unfortunately, despite the progress of modern surgical techniques, radical resection is possible only in l0%-25% of patients with CRC metastases confined to the liver.

Studies have suggested that DEB-IRI TACE may offer a novel approach to locoregional hepatic chemotherapy. DEB-IRI TACE allows a dose of irinotecan chemotherapy to be delivered directly into the liver, and thus has a significantly reduced side effect profile in comparison to systemic chemotherapy. It can be given alongside a reduced dose of systemic therapy or in some cases can be given instead of systemic therapies.

Pharmacokinetic analyses have shown the bioavailability from DC Bead (Biocompatibles UK, Farnham, United Kingdom)- based delivery of irinotecan is double that of intravenous infusion, attributable to reduced drug clearance for the former. Experimental animal studies have confirmed that DEB-IRI TACE induces lower early serum levels of irinotecan, a high and prolonged intratumoral level of irinotecan, and a greater rate of tumor necrosis compared with intraarterial or intravenous injection of irinotecan. Pilot clinical trials have suggested that DEB-IRI TACE administered in combination with systemic 5-fluorouracil and oxaliplatin in chemotherapy-naive patients or as a stand-alone regimen in patients with disease refractory to multiple lines of intravenous chemotherapy- may result in high rates of tumor response. In a randomized controlled study, DEB-IRI TACE showed a significant overall survival benefit with respect to a systemic regimen including irinotecan, 5-fluorouracil, and leucovorin in a series of 74 patients who had received at least two or three lines of chemotherapy.

Despite this initially promising evidence base, and a consensus document for treatment pathways, DEBIRI TACE use is not widespread.

This is partly due to a side effect profile, and partly due to a lack of standard technique or consensus.

There is a known side effect common to all forms of liver embolization, with or without the addition of chemotherapy or radiotherapy. The side effect profile is due to the mechanical effect of the device (beads) blocking small arteries within tumour tissue and normal liver tissue. The most common side effects and complications include pain and abscess formation due to embolic tissue ischaemia. These side effects are due to the device (DC Beads) rather than the addition of irinotecan chemotherapy.

A DEBIRI expert consensus meeting held in London in January 2017 suggested that UK practice varies very significantly between individual Trusts, despite a European consensus document which has suggested a defined treatment pathway. Only 2 of 12 UK centres had up to date retrospective information clarifying numbers of treatments, side effects, and length of hospital stay etc.

The greatest variations in individual practice was deemed to be three-fold

1. The number of treatments each patient receives.
2. The type of pain control given (General anaesthesia, sedo-analgesia, PCA pump, nerve block, or intra-arterial local anaesthetic).
3. The size and type of embolic bead.

These factors create a need for a registry to define current practice and analyse and compare individual and national variations within the centers already performing this procedure as a standard of care.

The registry would establish the varying national delivery techniques, complication profiles, quality of life, and health economic measures associated with delivery of the DC Bead device. This may help to determine causal associations between varying methods of device delivery and complication profiles and technical outcomes.

This is a prospective registry and service evaluation of current practice with respect to delivery of a CE marked device - DC Beads(BEBIRI).

The aim of the study is to:

1. Prospectively evaluate the number of centres providing DEBIRI
2. To determine the number of patients being treated nationally per year
3. To evaluate individual variations in practice with respect to number of treatments, method of pain control, side effect profile, and complication profile.
4. To collect patient specific data subsets to allow correlation and causal associations between these individual variations, and relate these to efficacy and survival during the study period.

The objectives are to assess current practice, to determine how well or poorly current practice correlates to published guidelines, and to determine which individual variations are associated with an increased complication profile.

The aim is to provide evidence to provoke reflection on individual variation in practice to assist the development of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Any race or sex
* Age 18-80.
* Histological diagnosis of Colorectal malignancy.
* Histological or radiological evidence of liver metastases from Colorectal Primary.
* Not suitable for surgical resection or ablation with curative intent.
* Metastatic liver burden occupying less than 50% of liver volume
* Liver dominant disease (defined as 80% or more of the overall whole body tumour burden confined to the liver).
* At least 1 measurable liver metastasis measuring over 1cm in size (RECIST 1.1 criteria to be applied).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1. ECOG 2 may occasionally be permissible on an individual patient by patient basis in line with local guidelines.
* Life expectancy 3+ months.
* Lack of pregnancy with ongoing use of acceptable contraceptive(in premenopausal women.
* Patent main portal vein.
* Adequate haematologic function as evidenced by: Haemoglobin of at least 8g/dl, platelets of at least 50 x 109/l, and International Normalised Ratio (INR) of under 1.5.
* Adequate liver function as evidence by a bilirubin level of less than twice the upper limit of normal.
* Deemed to be a suitable patient for DEBIRI treatment by MDT consensus.
* Consenting to inclusion in registry.

Exclusion Criteria:

* Any patient not fitting inclusion criteria.
* Previous or concurrent non-colorectal malignancy.
* No contraindication to Irinotecan administration.
* Uncorrectable clotting abnormality
* Documented allergy to contrast media that cannot be managed with standard care(steroids and antihistamines)
* Family, psychological, social or geographical circumstances preventing the patient from undergoing follow-up or from complying with protocol procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven colorectal carcinoma with synchronous or metachronous hepatic metastases selected for treatment with Irinotecan Drug-eluting beads.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Time to Hepatic Progression (TtHP) | 2 years after treatment
  Progression as measured by RECIST 1.1 criteria up to 2 years after treatment

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years after treatment
  Survival, defined as any time between start of treatment and death from any cause.
Adverse events | 4 months after treatment
  An adverse event (AE) is defined as any untoward or unfavourable medical occurrence, including any abnormal sign, symptom, or disease, temporally associated with the patient's participation in the research. It includes all adverse events regardless of seriousness or relatedness. A serious adverse event (SAE) is defined as an adverse event that: a. Results in death, b. Led to a serious deterioration in health that either: Results in a life-threatening illness or injury; results in a permanent impairment of a body structure or a body function; requires in-patient hospitalization or prolongation of existing hospitalization; results in medical or surgical intervention to prevent life threatening illness or injury; results in a persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, or, c. Led to fetal distress, foetal death or a congenital abnormality or birth defect
Quality of Life post DEBIRI delivery | 4 months after treatment
  Assessment of quality of life via The Edmonton Symptom Assessment System (ESAS).

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie Hospital NHS Foundation Trust, Manchester, United Kingdom